CLINICAL TRIAL: NCT05156281
Title: A Randomized, Double-blind, Double-dummy, Parallel-group Study, Comparing the Efficacy and Safety of Remibrutinib Versus Teriflunomide in Participants With Relapsing Multiple Sclerosis, Followed by Extended Treatment With Open-label Remibrutinib
Brief Title: Efficacy and Safety of Remibrutinib Compared to Teriflunomide in Participants With Relapsing Multiple Sclerosis (RMS)
Acronym: REMODEL-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLOU064C12302; 2023-509372-41-00 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: MS; RMS; RRMS; active secondary progressive multiple sclerosis SPMS; remibrutinib; LOU064; teriflunomide; adult; relapse; Expanded Disability Status Scale; T2 lesions; T1 lesions; GD- enhancing MRI; Neurofilament light chain; McDonald diagnostic criteria
MeSH Terms: conditions — Recurrence; Charcot-Marie-Tooth disease, Type 1F | interventions — remibrutinib; teriflunomide

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized in a 1:1 ratio
Who Masked: Participant, Investigator
Masking Description: In order to maintain blinding, a double-dummy design will be used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Remibrutinib - Core (Experimental): Remibrutinib tablet and matching placebo of teriflunomide capsule
  Interventions: Drug: Remibrutinib
- Teriflunomide - Core (Active Comparator): Teriflunomide capsule and matching placebo remibrutinib tablet
  Interventions: Drug: Teriflunomide
- Remibrutinib - Extension (Experimental): Participants on remibrutinib in Core will continue on remibrutinib tablet
  Interventions: Drug: Remibrutinib
- Remibrutinib - Extension (on teriflunomide in Core) (Experimental): Participants on teriflunomide in Core will switch to remibrutinib tablet
  Interventions: Drug: Remibrutinib

INTERVENTIONS:
Drug: Remibrutinib — tablet taken orally
  Other Names: LOU064
  Arms: Remibrutinib - Core; Remibrutinib - Extension; Remibrutinib - Extension (on teriflunomide in Core)
Drug: Teriflunomide — capsule taken orally
  Arms: Teriflunomide - Core

SUMMARY:
To compare the efficacy and safety of remibrutinib versus teriflunomide in patients with relapsing multiple sclerosis (RMS)

DETAILED DESCRIPTION:
The study CLOU064C12302 consists of an initial Core Part (CP) (maximum duration per participant of up to 30 months), followed by an Extension Part (EP, of up to 5 years duration) for eligible participants.

The Core Part is a randomized, double-blind, double-dummy, active comparator-controlled, fixed-dose, parallel-group, multi-center study in approximately 800 participants with relapsing multiple sclerosis (RMS).

The Extension Part is an open-label, single-arm, fixed-dose design in which eligible participants are treated with remibrutinib for up to 5 years.

A second study of identical design (CLOU064C12301) will be conducted simultaneously. Both studies will be conducted globally and data from the two studies will be pooled for some of the endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years of age
* Diagnosis of RMS according to the 2017 McDonald diagnostic criteria
* At least: 1 documented relapse within the previous year. OR 2 documented relapses within the previous 2 years, OR 1 active Gadolinium (Gd)-enhancing lesion in the 12 months.
* EDSS score of 0 to 5.5 (inclusive)
* Neurologically stable within 1 month

Exclusion Criteria:

* Diagnosis of primary progressive multiple sclerosis (PPMS)
* Disease duration of more than 10 years in participants with EDSS score of 2 or less at screening
* History of clinically significant CNS disease other than MS
* Ongoing substance abuse (drug or alcohol)
* History of malignancy of any organ system (other than complete resection of localized basal cell carcinoma of the skin or in situ cervical cancer),
* Participants with history of confirmed Progressive Multifocal Leukoencephalopathy (PML) or Neurological symptoms consistent with PML
* suicidal ideation or behavior
* Evidence of clinically significant cardiovascular, neurological, psychiatric, pulmonary , renal, hepatic, endocrine, metabolic, hematological disorders or gastrointestinal disease that can interfere with interpretation of the study results or protocol adherence
* Participants who have had a splenectomy
* Active clinically significant systemic bacterial, viral, parasitic or fungal infections
* Positive results for syphilis or tuberculosis testing
* Uncontrolled disease states, such as asthma, or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids
* Active, chronic disease of the immune system (including stable disease treated with immune therapy (e.g. Leflunomide, Methotrexate)) other than MS (e.g. rheumatoid arthritis, systemic lupus erythematosus, etc.) with the exception of well-controlled diabetes or thyroid disorder.
* Participants with a known immunodeficiency syndrome (AIDS, hereditary immune deficiency, drug induced immune deficiency), or tested positive for HIV antibody
* History or current treatment for hepatic disease including but not limited to acute or chronic hepatitis, cirrhosis (including all Child-Pugh classes) or hepatic failure or any chronic liver or biliary disease.
* History of severe renal disease or creatinine level
* Participants at risk of developing or having reactivation of hepatitis
* Hematology parameters at screening:

  * Hemoglobin: < 10 g/dl (<100g/L)
  * Platelets: < 100000/mm3 (<100 x 109/L)
  * Absolute lymphocyte count < 800/mm3 (<0.8 x 109/L)
  * White blood cells: <3 000/mm3 (<3.0 x 109/L)
  * Neutrophils: < 1 500/mm3 (<1.5 x 109/L)
  * B-cell count < 50% lower limit of normal (LLN) or total IgG & total IgM < LLN (only required for participants who had a history of receiving B-cell therapies, such as rituximab, ocrelizumab or ofatumumab, prior to screening)
* History or current diagnosis of significant ECG abnormalities
* Resting QTcF ≥450 msec (male) or ≥460 msec (female) at pre-treatment as per central ECG reading at screening visit
* Use of other investigational drugs
* Requirement for anticoagulant medication or use of dual anti-platelet therapy Significant bleeding risk or coagulation disorders,
* History of gastrointestinal bleeding
* Major surgery within 8 weeks prior to screening
* History of hypersensitivity to any of the study drugs or excipients
* Pregnant or nursing (lactating) female participants, prior to randomization
* Women of childbearing potential not using highly effective contraception
* Sexually active males not agreeing to use condom
* Have received any live or live-attenuated vaccines within 6 weeks of randomization or requirement to receive these vaccinations during study
* Use of strong CYP3A4 inhibitors or use of moderate or strong CYP3A4 inducers within two weeks prior to randomization

Inclusion to Extension part:

• Participants who complete the Core Part of the study on double-blind study treatment and conduct the Accelerated Elimination Procedure (AEP)

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1011 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Annualized relapse rate (ARR) of confirmed relapses [Core Part] | From Baseline, up to 30 months
  ARR is the average number of confirmed MS relapses in a year

SECONDARY OUTCOMES:
Time to 3-month confirmed disability progression (3mCDP) on Expanded Disability Status Scale (EDSS) [Core Part] (pooled data) | Baseline up to 30 months
  Time to 3-month confirmed disability progression (3mCDP) is defined as an increase in Expanded Disability Status Scale (EDSS) which is sustained for at least 3 months
Time to 6-month confirmed disability progression (6mCDP) on EDSS [Core Part] (pooled data) | Baseline up to 30 months
  Time to 6-month confirmed disability progression (6mCDP) is defined as an increase in Expanded Disability Status Scale (EDSS) which is sustained for at least 6 months
Annualized rate of new or enlarging T2 lesion [Core Part] | Baseline up to 30 months
  Number of new/newly enlarged T2 lesions per year
Neurofilament light chain (Nfl) [Core Part] | Baseline up to 30 months
  Neurofilament light chain (NfL) concentration in serum
Number of Gd-enhancing T1 lesions per MRI scan [Core Part] | Baseline up to 30 months
  Average number of Gd-enhancing T1 lesions per scan
Percentage of participants with No Evidence of Disease Activity-3 (NEDA-3) [Core Part] (pooled data) | Baseline up to 30 months
  Percentage of participants with No Evidence of Disease Activity-3 (NEDA-3), as assessed by absence of confirmed MS relapses, 6mCDP and new/enlarging T2 lesions on MRI
Time to first confirmed relapse [Core Part] | Baseline up to 30 months
  Change in the Expanded Disability Status Scale (EDSS), an increase of at least 0.5 points on the EDSS (total) score, or an increase of at least 1 point on at least two functional scores (FSs), or an increase of at least 2 points on at least one FS, excluding changes involving bowel/bladder or cerebral FS, compared to the previous available rating.
Time to 6-month confirmed disability improvement (6mCDI) on EDSS [Core Part] (pooled data) | Baseline up to 30 months
  Decrease in Expanded Disability Status Scale Score (EDSS) which is sustained for at least 6 months
Time to 3-months confirmed disability progression (3mCDP) and 6-month confirmed disability progression (6mCDP) independent of relapse activity (PIRA) [Core Part] (pooled data) | Baseline up to 30 months
  Time to 3-month confirmed disability progression (3mCDP) and 6-month confirmed disability progression (6mCDP) is defined as an increase in Expanded Disability Status Scale (EDSS) which is sustained for at least 3 months or 6 months, respectively, without an on-study relapse before or on the day of a progression eve
Change from baseline in the Symbol Digit Modalities Test (SDMT) [Core Part] (pooled data) | Baseline up to 30 months
  Symbol Digit Modalities Test (SDMT), an array of symbols paired with empty spaces, measures processing in speed; participants verbally match the number for each symbol as rapidly as possible. The score is the number of correctly coded items in 90 seconds. Higher scores indicate improvement. Lower scores indicate worsening
Time to 6-month confirmed worsening by at least 20% in the Timed 25-foot walk test (T25FW) [Core Part] (pooled data) | Baseline, up to 30 months
  The patient walking speed to cover 25-foot distance is recorded in seconds. Longer time indicates poorer lower limb function. 20% worsening is defined as 20% increase from baseline T25FW score
Time to 6-month confirmed worsening by at least 20% in the Timed 9-hole peg test (9HPT) (pooled data) [Core Part] (pooled data) | Baseline up to 30 months
  The patient's right and left arm function to peg 9 holes measured in seconds. Longer time indicates poorer upper limb function. 20% worsening is defined as 20% increase from baseline 9HPT score in at least one hand (average of two trials per hand)
Time to composite 6-month confirmed disability Progression (CDP) [Core Part] (pooled data) | Baseline up to 30 months
  The composite involves CDP and worsening by at least 20% in T25FW and 9HPT
Change from Baseline in T2 lesion volume [Core Part] | Baseline up to 30 months
  Change from baseline in total T2 lesion volume.
Change from baseline in Multiple Sclerosis Impact Scale (MSIS-29) [Core Part] | Baseline up to 30 months
  29-item, self-administered questionnaire that includes 2 domains, physical and psychological. Responses are captured on a 4-point scale ranging from "not at all" (1) to "extremely" (4), where higher scores reflect greater impact on day to day life
Number of participants with Adverse events and Serious adverse events(SAE) [Core Part] | Baseline up to 30 months
  Adverse events and SAEs including clinically significant, laboratory data, vital signs, electrocardiogram (ECG), Columbia Suicide Severity Rating
Pharmacokinetics of remibrutinib [Core Part] | Month 1, Month 6
  Blood concentrations of remibrutinib
Number of participants with Adverse events and Serious adverse events (SAE) [Extension Part] | Day 1 Extension up to 5 years
  Adverse events and SAEs including clinically significant, laboratory data, vital signs, electrocardiogram (ECG), Columbia Suicide Severity Rating
Annualized relapse rate (ARR) of confirmed relapses [Extension Part] | Day 1 Extension up to 5 years
  ARR is the average number of confirmed MS relapses in a year
Annualized rate of new or enlarging T2 lesion [Extension Part] | Day 1 Extension up to 5 years
  Number of new/newly enlarged T2 lesions per year
Time to 6-month confirmed disability progression (6mCDP) on EDSS [Extension Part] | Day 1 Extension up to 5 years
  Time to 6-month confirmed disability progression (6mCDP) is defined as an increase in Expanded Disability Status Scale (EDSS) which is sustained for at least 6 months
Change from baseline in the Symbol Digit Modalities Test (SDMT) [Extension Part] | Day 1 Extension up to 5 years
  Symbol Digit Modalities Test (SDMT), an array of symbols paired with empty spaces, measures processing in speed; participants verbally match the number for each symbol as rapidly as possible. The score is the number of correctly coded items in 90 seconds. Higher scores indicate improvement. Lower scores indicate worsening
Neurofilament light chain (NfL) [Extension Part] | Day 1 Extension up to 5 years
  Neurofilament light chain (NfL) concentration in serum
Change from baseline in Multiple Sclerosis Impact Scale (MSIS-29) [Extension Part] | Day 1 Extension up to 5 years
  29-item, self-administered questionnaire that includes 2 domains, physical and psychological. Responses are captured on a 4-point scale ranging from "not at all" (1) to "extremely" (4), where higher scores reflect greater impact on day to day life

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (208):
- United States (53):
  - Ctr for Neurology and Spine, Phoenix, Arizona
  - Vladimir Royter MD APMC, Hanford, California
  - VA Greater LA Healthcare System, Los Angeles, California
  - Regina Berkovich MD PhD Inc, West Hollywood, California
  - CU Anschutz Med Campus, Aurora, Colorado
  - Colorado Neurological Research PC, Denver, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Georgetown University Hospital Research, Washington D.C., District of Columbia
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Nova Clinical Research LLC, Bradenton, Florida
  - University of Florida, Gainesville, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Neurology Associates PA, Maitland, Florida
  - Gables Neurology, Miami, Florida
  - UM Department Of Neurology, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Advent Health Orlando, Orlando, Florida
  - Humanity Clinical Research, Pembroke Pines, Florida
  - Emerald Coast Neurology, Pensacola, Florida
  - Brain and Spine Institute, Port Orange, Florida
  - Vero Beach Neurology, Vero Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Methodist Neuroscience Institute, Merrillville, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - Baptist Physicians Lexington, Nicholasville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Clinre Comprehensive Neurology, Frederick, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Kansas City VA Medical Center, Kansas City, Missouri
  - South Shore Neurologic Associates, Patchogue, New York
  - True North Neurology, Port Jefferson, New York
  - University Of NC At Chapel Hill, Chapel Hill, North Carolina
  - Piedmont HealthCare, Charlotte, North Carolina
  - The Boster Ctr for MS, Columbus, Ohio
  - Neurology Diagnostics Inc, Dayton, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Medical Uni of South Carolina, Charleston, South Carolina
  - Premier Neurology, Greenville, South Carolina
  - Metrolina Neurological Associates PA, Old Point Station, South Carolina
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Neurology Consultants Of Dallas PA, Dallas, Texas
  - Med Research Inc, El Paso, Texas
  - Lone Star Neurology, Frisco, Texas
  - UT Health MARC Medical Arts and Research Center, San Antonio, Texas
  - Lonestar Neurology of San Antonio, San Antonio, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - Baylor Scott and White, Temple, Texas
  - Virginia Mason Medical Centre, Seattle, Washington
  - University of Washington MS Clinic, Seattle, Washington
  - Elligo Health Research, Crab Orchard, West Virginia
  - Ascension St Francis Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (6):
  - Novartis Investigative Site, Bombal, Mendoza Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Córdoba
- Brazil (6):
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Joinville, Santa Catarina
  - Novartis Investigative Site, São Paulo
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (8):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saint-Jérôme, Quebec
- China (8):
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Yinchuan, Ningxia
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Croatia (4):
  - Novartis Investigative Site, Split, HRV
  - Novartis Investigative Site, Varaždin, HRV
  - Novartis Investigative Site, Vukovar
  - Novartis Investigative Site, Zagreb
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Teplice
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- France (13):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Gonesse
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Poissy
  - Novartis Investigative Site, Toulouse
- Germany (3):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
- Greece (5):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chaïdári
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Larissa
  - Novartis Investigative Site, Thessaloniki
- India (7):
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Amritsar, Punjab
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Kolkata, West Bengal
- Italy (8):
  - Novartis Investigative Site, Brindisi, BR
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Napoli
- Japan (20):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Ichihara, Chiba
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Moriguchi, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Higashi-Matsuyama, Saitama
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Kobe
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Niigata
- Mexico (4):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Chihuahua City
  - Novartis Investigative Site, Mexico City
  - Novartis Investigative Site, Querétaro
- Poland (7):
  - Novartis Investigative Site, Plewiska, Poznan
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Glogow Wielkopolski
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zabrze
- Portugal (6):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Santa Maria da Feira
- Caribbean Center for Clinical Research, Inc, Guaynabo, Puerto Rico
- Romania (4):
  - Novartis Investigative Site, Brasov, ROM
  - Novartis Investigative Site, Constanța, ROM
  - Novartis Investigative Site, Campulung Muscel
  - Novartis Investigative Site, Constanța
- Slovakia (2):
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
- Slovenia (3):
  - Novartis Investigative Site, Celje
  - Novartis Investigative Site, Ljubljana
  - Novartis Investigative Site, Maribor
- South Africa (3):
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Pretoria
  - Novartis Investigative Site, Rosebank
- Spain (16):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Vitoria-Gasteiz, Araba
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Albacete, Castille-La Mancha
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Logroño, La Rioja
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Torrejón de Ardoz, Madrid
  - Novartis Investigative Site, Gijón, Principality of Asturias
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Lleida
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Stockholm, Sweden
- Turkey (Türkiye) (10):
  - Novartis Investigative Site, Samsun, Atakum
  - Novartis Investigative Site, Izmir, Balcova
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Izmir, Karabaglar
  - Novartis Investigative Site, Kayseri, Melikgazi
  - Novartis Investigative Site, Bursa, Nilufer
  - Novartis Investigative Site, Istanbul, Pendik
  - Novartis Investigative Site, Istanbul, Sancaktepe
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Konya
- United Kingdom (3):
  - Novartis Investigative Site, Inverness, Invernesshire
  - Novartis Investigative Site, Canterbury, Kent
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com